CLINICAL TRIAL: NCT00593632
Title: A Controlled Trial of High Dietary Fiber Intake on Serum Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Attune Foods (Unknown)
Responsible Party: Principal Investigator, Wael Jaber, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-852
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Hyperlipidemia
Keywords: low HDL
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Fiber Intake (Experimental): Two 3/4 Cup servings of high fiber Uncle Sam cereal daily
  Interventions: Dietary Supplement: Uncle Sam Cereal

INTERVENTIONS:
Dietary Supplement: Uncle Sam Cereal — two 3/4 cup servings daily of Uncle Sam Cereal dietary instruction on high fiber diet

SUMMARY:
The study evaluates high fiber diet intake in patients with hyperlipidemia.

DETAILED DESCRIPTION:
Dietary fiber intake has been shown to have modest effect in lowering cholesterol. However, most of these studies were done with 20g/daily fiber intake. Not much is known about high dietary fiber intake (30-40 g/day) and serum cholesterol. Also, there have been small studies that have shown modest decrease in oxidative stress by increasing dietary fiber intake. The goal of our study is to determine the efficacy /safety of high dietary fiber intake in raising HDL, lowering LDL, and lowering oxidative stress in patients with hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

* All primary and secondary prevention patients aged 18 to 80 years with known or newly diagnosed isolated hypercholesteremia or combined hyperlipidemia.
* Inclusion criteria include patients with HDL < 35 mg/dL for a man or < 45mg/dL for women irrespective of LDL level.

Exclusion Criteria:

* Any patients with unstable angina, untreated hypothyroidism, uncontrolled diabetes, other endocrine or metabolic diseases not actively treated, acute inflammatory diseases, severe gastrointestinal diseases, chronic renal insufficiency (GFR<30), end stage renal disease, liver disease or other severe diseases such as cancer, triglyceride level greater than 600 mg/dL, pregnant females, chronic use of systemic corticosteroid, or anticoagulants.
* Patients who were recently started or recently had their lipid lowering medications changed within the last 4 weeks will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To test whether 30-40g of daily dietary fiber increases HDL, lowers total cholesterol and LDL levels in patients at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
To test whether Lipoprotein (a), triglyceride level, LDL: HDL ratio, fibrinogen, CRP, Urine f1 2 isoprostane and body weight will be lowered in patients after 12weeks. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wael A Jaber, MD, Principal Investigator — The Cleveland Clinic; Leslie Cho, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No